CLINICAL TRIAL: NCT02908256
Title: Randomized Double-blind Comparison of Intraoperative Volume Replacement Determined by the Plethysmograph Variability Index (PVI) With That Determined by the Delta PP in the Digestive, Gynecological, Urological, and Abdominal Surgery and Their Impact on the Length of Stay
Brief Title: Comparison of Intraoperative Volume Replacement Determined by the Plethysmograph Variability Index (PVI) With That Determined by the Delta PP in the Digestive, Gynecological, Urological, and Abdominal Surgery and Their Impact on the Length of Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Philippe VAN DER LINDEN, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUB-GIFA
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Abdomino-pelvic Surgery
Keywords: PVI; delta PP; vascular filling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI group (Experimental): Monitoring of the PVI during the surgical intervention
  Interventions: Drug: Geloplasma (PVI)
- Delta PP group (Active Comparator): Monitoring of the deltaPP during the surgical intervention
  Interventions: Drug: Geloplasma (delta PP)

INTERVENTIONS:
Drug: Geloplasma (PVI) — In the PVI group, a filling solution (geloplasma) will be given as a bolus of 250 ml administered in 10 minutes if the PVI>15% during more than 5 minutes. The bolus will be repeated if the PVI remains over 15%.
  Arms: PVI group
Drug: Geloplasma (delta PP) — In the delta PP group, a filling solution (geloplasma) will be given as a bolus of 250 ml administered in 10 minutes if the delta PP> 13% during more than 5 minutes. The bolus will be repeated if the delta PP remains over 13%.
  Arms: Delta PP group

SUMMARY:
An optimal intraoperative fluid replacement reduces the hospital stay, the admissions in the intensive care unit and the mortality rate after a major surgery.

Different criteria are used to guide the optimal vascular filling of a patient. Among the various monitoring for the last twenty years are parameters originating from the respiratory variations of the arterial pressure curves and the pulse oximetry.

On arterial curves, the Systolic Pressure Variation (SPV) is the difference between the maximum systolic pressure (DeltaUp) and the minimal one (DeltaDown).On the oxygen saturometry curves obtained with the Masimo Radical7, the plethysmographic variability index (PVI) corresponds to the formula (PImax-PImin/PImax X 100%) where PI corresponds to the quotient expressed in % between the pulsed infrared absorption signal and the continuous absorption signal.

It has been demonstrated that the dynamic indexes were better than the static indexes to determine the response to the vascular filling. A meta-analysis showed that the dynamic changes of the variables derived from the arterial pressure curve of patients under mechanic ventilation could predict the vascular filling responsiveness with a high specificity and sensibility. The same thing applies to the variables derived from the pulsed oxymetry curves.

Furthermore, monitoring and minimizing, through the vascular filling, the variations of the pulsated arterial pressure (delta PP) induced by the mechanic ventilation during a high risk surgery allows to reduce the postoperative complications and the hospital length of stay. This has not yet been proved for the non invasive parameters (IP and PVI).

The goal of this study is thus to compare a non invasive strategy (based on PVI) to an invasive strategy (based on the deltaPP) of perioperatory filling during abdomino-pelvic interventions (digestive, gynecologic, urologic), in order to test their equivalence and measure their impact in terms of hospital stay.

This record is linked to the NCT02709252 record and share the same cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal-pelvic surgery (digestive, gynecologic, urologic) with laparotomy or laparoscopy
* Surgery duration superior to 1 hour

Exclusion Criteria:

* ASA score of 4
* BMI > 35
* supraventricular arrythmia (isolated extrasystoles excepted)
* cardiac insufficiency (F.E < 25 %)
* severe peripheric vascular affections
* severe respiratory affections
* terminal renal insufficiency (creatine clear and < 30 mL/min)
* gelatin allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | average of 5 days

SECONDARY OUTCOMES:
EVA score | up to 72 hours
  post surgery pain scoring
number of anti-emetics administered | up to 72 hours
length of stay in recovery room | up to 24 hours
First time up | up to 72 hours
  First time up/ first time sitting in a chair

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van Der Linden, MD, Principal Investigator — CHU Brugmann

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bundgaard-Nielsen M, Holte K, Secher NH, Kehlet H. Monitoring of peri-operative fluid administration by individualized goal-directed therapy. Acta Anaesthesiol Scand. 2007 Mar;51(3):331-40. doi: 10.1111/j.1399-6576.2006.01221.x. PMID 17390421
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Cannesson M, Desebbe O, Rosamel P, Delannoy B, Robin J, Bastien O, Lehot JJ. Pleth variability index to monitor the respiratory variations in the pulse oximeter plethysmographic waveform amplitude and predict fluid responsiveness in the operating theatre. Br J Anaesth. 2008 Aug;101(2):200-6. doi: 10.1093/bja/aen133. Epub 2008 Jun 2. PMID 18522935
- [Background] Zimmermann M, Feibicke T, Keyl C, Prasser C, Moritz S, Graf BM, Wiesenack C. Accuracy of stroke volume variation compared with pleth variability index to predict fluid responsiveness in mechanically ventilated patients undergoing major surgery. Eur J Anaesthesiol. 2010 Jun;27(6):555-61. doi: 10.1097/EJA.0b013e328335fbd1. PMID 20035228
- [Background] Michard F, Lopes MR, Auler JO Jr. Pulse pressure variation: beyond the fluid management of patients with shock. Crit Care. 2007;11(3):131. doi: 10.1186/cc5905. PMID 17521454
- [Derived] Coeckelenbergh S, Delaporte A, Ghoundiwal D, Bidgoli J, Fils JF, Schmartz D, Van der Linden P. Pleth variability index versus pulse pressure variation for intraoperative goal-directed fluid therapy in patients undergoing low-to-moderate risk abdominal surgery: a randomized controlled trial. BMC Anesthesiol. 2019 Mar 9;19(1):34. doi: 10.1186/s12871-019-0707-9. PMID 30851740